CLINICAL TRIAL: NCT06949618
Title: Feasibility and Effectiveness of Repetitive Transcranial Magnetic Stimulation in Patients With Cancer Pain
Brief Title: Repetitive Transcranial Magnetic Stimulation in Cancer Pain Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202209046
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Pain; Cancer
MeSH Terms: conditions — Pain; Neoplasms | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Repetitive transcranial magnetic stimulation (Experimental)
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- Sham Repetitive transcranial magnetic stimulation (Sham Comparator)
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — Repetitive transcranial magnetic stimulation toward for cancer pain (real and sham control)

SUMMARY:
Over half of cancer patients experience cancer-related pain. Despite advances in pain management with opioids, many patients continue to suffer from chronic cancer pain. The underlying mechanisms of cancer-related pain remain poorly understood, but they may be linked to brain neuroplasticity. As a result, some researchers suggest that targeting the motor cortex in cancer patients could improve pain management. However, few studies have investigated the effectiveness of remodeling neuroplasticity with repetitive transcranial magnetic stimulation (rTMS) to reduce cancer-related pain. To validate the use of rTMS in cancer-related pain, we plan to conduct a randomized controlled trial involving 30 cancer pain patients. Participants will be randomly assigned to receive either rTMS or sham rTMS treatment. Functional magnetic resonance imaging (fMRI) and pain index assessments will be conducted before and after the treatment to evaluate the outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have cancer pain symptoms, confirmed by a physician as cancer pain or neuropathic cancer pain
2. Experienced the worst pain NRS score ≥ 4
3. The patient demonstrate good cognition and is able to cooperate with the assessment of pain severity.
4. The estimated survival time exceeds 3 months.
5. Pre-existing bisphosphonate, chemotherapy, and hormonal therapy regimens remained unchanged throughout the study.

Exclusion Criteria:

1. Individuals who have undergone head surgery or have metal implants in the head.
2. Individuals with implanted cardiac pacemakers or cochlear prostheses.
3. Have a history of epilepsy.
4. Patients diagnosed with primary brain tumors or metastatic brain lesions.
5. Present with additional neurological, psychiatric, or severe medical disorders.
6. Individuals with metallic implants located in the cranial or cervical regions.
7. Women who are pregnant.
8. Presence of acute pain in any body region attributable to other medical conditions. -

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2026-12-16 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory, BPI | Assess the BPI outcome before the intervention, after 1 week and 2 weeks of intervention, as well as 1 week and 4 weeks after the intervention is completed.
  BPI is to assess the severity of pain and the impact of pain on daily functions, including Severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours.
McGill Pain Questionnaire | Assess MPQ scores before the intervention, after 1 week and 2 weeks of intervention, as well as 1 week and 4 weeks after the intervention is completed.
  The McGill Pain Questionnaire (MPQ) is a self-report measure used by patients with various diagnoses to assess pain. It consists of 78 words, from which respondents select those that best describe their pain experience. The words are categorized as follows:
  Dimensions 1 to 10 (pain descriptors): 3 words
  Dimensions 11 to 15 (affective components of pain): 3 words
  Dimension 16 (evaluation of pain): 1 word
  Dimensions 17 to 20 (miscellaneous): 1 word.
  Scores are calculated by summing the values associated with each selected word, with scores ranging from 0 (no pain) to 78 (severe pain). Qualitative differences in pain are reflected in the respondent's word choices.

SECONDARY OUTCOMES:
Numerical Rating Scale, NRS | Assess the NRS scale before the intervention, after 1 week and 2 weeks of intervention, as well as 1 week and 4 weeks after the intervention is completed.
  The Numeric Rating Scale (NRS) is commonly used to measure pain intensity and is well validated. It is scored from 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable
Visual Analogue Scale , VAS | Assess the VAS scale before the intervention, after 1 week and 2 weeks of intervention, as well as 1 week and 4 weeks after the intervention is completed.
  The Visual Analog Scale (VAS) is a validated, subjective measure of both acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum from 'no pain' to 'worst pain.'
Resting-state functional imaging, rsfMRI | Assess the fMRI results before the intervention and after 2 weeks of interventions.
  In fMRI, by adding each pixel, the time course of a pixel is related to the average time course of the corresponding region of interest (ROI). In this context, the cross-correlation coefficient map for each seed ROI will be generated. This cross-correlation coefficient map will then undergo Fisher's z-transformation to approximate a normal distribution.
Beck Depression Inventory, BDI | Assess the BDI scale before the intervention, after 1 week and 2 weeks of intervention, as well as 1 week and 4 weeks after the intervention is completed.
  BDI is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Each answer is being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.
The 36-Item Short Form Survey quality of life | Assess the The SF-36 outcome before the intervention, after 1 week and 2 weeks of intervention, as well as 1 week and 4 weeks after the intervention is completed.
  The 36-Item Short Form Survey (It comprises 36 questions that cover eight domains of health) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. It comprises 36 questions that cover eight domains of health.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No